CLINICAL TRIAL: NCT00857311
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Probe Study With an Additional Open-Label Control Arm to Evaluate the Safety and Immunogenicity of a 3-Dose Regimen of the MRKAd5 HIV-1 Gag Vaccine in Subjects With Chronic Hepatitis C Virus Infection
Brief Title: MRKAd5 HIV-1 Gag Vaccine (V520) in Subjects With Chronic Hepatitis C (V520-022) (COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V520-022; 2009_556
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MRKAd5 HIV-1 gag vaccine 1x10^9 vp/dose (Experimental): Participants administered MRKAd5 HIV-1 gag vaccine 1x10^9 viral particles (vp)/dose (V520), on Day 1, Week 4, and Week 26.
  Interventions: Biological: MRKAd5 HIV-1 gag vaccine (V520)
- MRKAd5 HIV-1 gag vaccine 1x10^10 vp/dose (Experimental): Participants were to be administered MRKAd5 HIV-1 gag 1x10^10 vp/dose (V520) on Day 1, Week 4, and Week 26.
  Per a letter dated 30-Aug-2005 all sites were notified that due to recruitment challenges enrollment would be halted as of 01-Oct-2005. Consequently, no participants were enrolled in the group MRKAd5 HIV-1 gag 1x10^10 vp/dose.
  Interventions: Biological: MRKAd5 HIV-1 gag vaccine (V520)
- Placebo (Experimental): Participants administered placebo to MRKAd5 HIV-1 gag vaccine (V520) on Day 1, Week 4, and Week 26.
  Interventions: Biological: Comparator: Placebo
- Open Label Tetanus and Diptheria Toxoids Adsorbed (Sham Comparator): Participants were to be administered open label tetanus and diptheria toxoids adsorbed (Td) at Day 1 only.
  Per a letter dated 30-Aug-2005 all sites were notified that due to recruitment challenges enrollment would be halted as of 01-Oct-2005. Consequently, no participants were enrolled in this group.
  Interventions: Biological: Comparator: Open Label Tetanus and Diptheria Toxoids Adsorbed

INTERVENTIONS:
Biological: MRKAd5 HIV-1 gag vaccine (V520) — 3-dose prime boosting regimen of 1.0-mL intramuscular injections of 1x10^9 viral particles/dose of MRKAd5 HIV-1 gag vaccine (V520) at Day 1 and Weeks 4 and 26
  Arms: MRKAd5 HIV-1 gag vaccine 1x10^9 vp/dose
Biological: Comparator: Placebo — 1.0 mL intramuscular injection of Placebo at Day 1 and Weeks 4 and 26
  Arms: Placebo
Biological: Comparator: Open Label Tetanus and Diptheria Toxoids Adsorbed — 0.5 mL Open Label Tetanus and Diptheria Toxoids Adsorbed (Td) intramuscular injection at Day 1 only
  Arms: Open Label Tetanus and Diptheria Toxoids Adsorbed
Biological: MRKAd5 HIV-1 gag vaccine (V520) — 3-dose prime boosting regimen of 1.0-mL intramuscular injections of 1x10^10 viral particles/dose of MRKAd5 HIV-1 gag vaccine (V520) at Day 1 and Weeks 4 and 26
  Arms: MRKAd5 HIV-1 gag vaccine 1x10^10 vp/dose

SUMMARY:
A Study to assess the general safety and tolerability of the administration of a 3-dose prime/boost regimen of the MRKAd5 HIV-1 gag vaccine (V520) in subjects with chronic hepatitis C virus infection.

ELIGIBILITY:
Inclusion Criteria:

* Subject who is of reproductive potential agrees to use a acceptable method of birth control through week 52 of the study

Exclusion Criteria:

* Subject weighs less than 110 lbs.
* Subject has received treatment for hepatitis C virus infection in the 3 months before enrollment in this study or is anticipated to begin treatment with in 1 year after enrollment
* Subject has any history of anaphylaxis or allergy to vaccine components
* Subject has any history of anaphylaxis or allergy to Tetanus and Diphtheria Toxoids Adsorbed (Td)
* Subject has clinical signs suggestive of cirrhosis
* Subject has had a liver biopsy showing bridging fibrosis or cirrhosis
* Subject is HBsAg positive
* Subject has other known chronic liver disease
* Subject has evidence of hepatocellular carcinoma on liver biopsy
* Subject has had a liver transplant or is anticipated to have a liver transplant within 1 year of enrollment
* Subject has been vaccinated with a live virus vaccine in the past 30 days
* Subject has been vaccinated with an inactive virus vaccine in the past 14 days
* Female subject is pregnant or breast-feeding, Male subject is planning to impregnate
* Subject has active drug or alcohol abuse
* Subject is at high risk for HIV infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2004-05; Primary Completion 2006-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants had to be at low risk of acquiring human immunodeficiency virus (HIV) infection, and had to meet a number of laboratory criteria. They could not have received treatment for hepatitis C virus infection in the 3 months prior to enrollment and must not anticipate to begin treatment with in 1 year after enrollment.
Period: Overall Study
Arm/Group | MRKAd5 HIV-1 Gag Vaccine 1x10^9 vp/Dose | MRKAd5 HIV-1 Gag Vaccine 1x10^10 vp/Dose | Placebo | Open Label Tetanus and Diptheria Toxoids Adsorbed
Started | 9 | 0 | 8 | 0
Completed | 8 | 0 | 8 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MRKAd5 HIV-1 Gag Vaccine 1x10^9 vp/Dose | MRKAd5 HIV-1 Gag Vaccine 1x10^10 vp/Dose | Placebo | Open Label Tetanus and Diptheria Toxoids Adsorbed | Total
Number analyzed (Participants) | 9 | 0 | 8 | 0 | 17
Age, Customized [Mean (Full Range); unit: years] | 41.4 [33 to 54] |  | 39.3 [22 to 49] |  | 40.4 [22 to 54]
Gender [Number; unit: participants]
  Female | 5 |  | 4 |  | 9
  Male | 4 |  | 4 |  | 8
Region of Enrollment [Number; unit: participants]
  United States | 9 |  | 8 |  | 17

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Systemic and Laboratory Adverse Events (AE)
Description: Adverse experiences collected include serious and non serious systemic AEs, injection-site AEs, and laboratory AEs. Systemic and laboratory AEs include any unfavorable & unintended change in the structure, function, or chemistry of the body. Injection-site AEs include any swelling, redness, pain or tenderness at the injection site. All injection site AEs were collected up to 5 days after any vaccine dose.
Time Frame: up to Week 260 (234 weeks after boost injection) for systemic AEs, 29 days after any dose for laboratory AEs, and 5 days after any dose for injection-site AEs
Measure: Number; unit: Participants
Arm/Group | MRKAd5 HIV-1 Gag Vaccine 1x10^9 vp/Dose | Placebo
Number analyzed (Participants) | 9 | 8
Participants
  With non-serious systemic AEs | 8 | 6
  With serious systemic AEs | 2 | 2
  With non-serious injection-site AEs | 3 | 1
  With serious injection-site AEs | 0 | 0
  With non-serious laboratory AEs | 4 | 1
  With serious laboratory AEs | 0 | 0

2. Secondary Outcome: Immune Response by Levels of Unfractionated Gag-specific IFN-gamma Following a 3-dose Vaccine Regimen
Description: Participants expressing HIV antigens (gag) secrete antigen specific interferon-gamma (IFN-gamma). Levels of unfractionated gag-specific IFN-gamma were to be measured using an Enzyme Linked Immunospot Assay (ELISPOT), which measures spot forming cells per 10^6 peripheral blood mononuclear cells (SFC per million PBMCs).
  No immunogenicity analyses were performed because the results from a previous study, V520-023 (NCT00095576), which used the same vaccine as the one used in this study (NCT00857311) proved it was not efficacious.
Time Frame: Week 30 (4 weeks after boost injection)
Population: No analysis was performed.
Arm/Group | MRKAd5 HIV-1 Gag Vaccine 1x10^9 vp/Dose | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Participants With Vaccine-related Clinical (Systemic and Injection-site), and Laboratory Adverse Events (AE)
Description: Serious and non serious clinical (systemic and injection-site AEs), and laboratory AEs were collected. Systemic and laboratory AEs reflect any unfavorable & unintended change in the structure, function, or chemistry of the body. Injection-site AEs include any swelling, redness, pain or tenderness at the injection site.
  Vaccine-related AEs are those determined by the investigator to be possibly, probably, or definitely related to the administration of the vaccine.
Time Frame: up to Week 78 (52 weeks after boost injection) for systemic AEs, 29 days after any dose for laboratory AEs, and 5 days after any dose for injection-site AEs
Measure: Number; unit: Participants
Arm/Group | MRKAd5 HIV-1 Gag Vaccine 1x10^9 vp/Dose | Placebo
Number analyzed (Participants) | 9 | 8
Participants
  With non-serious vaccine-related (VR) clinical AEs | 5 | 1
  ---With non-serious VR systemic AEs | 3 | 1
  ---With non-serious VR injection-site AEs | 3 | 1
  With serious VR clinical AEs | 0 | 0
  ---With serious VR systemic AEs | 0 | 0
  ---With serious VR injection-site AEs | 0 | 0
  With non-serious VR laboratory AEs | 2 | 0
  With serious VR laboratory AEs | 0 | 0
  discontinued due to non-serious VR clinical AE | 0 | 0
  discontinued due to serious VR clinical AE | 0 | 0
  discontinued due to VR non-serious laboratory AE | 0 | 0
  discontinued due to VR serious laboratory AE | 0 | 0

ADVERSE EVENTS:
Time Frame: Injection-site AEs up to 5 days after vaccination, non-serious systemic AEs and laboratory AEs up to 29 days after vaccination, serious AEs for the entire study period (Week 260).
Arm/Group | MRKAd5 HIV-1 Gag Vaccine 1x10^9 vp/Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 2/9 | 2/8
Other Adverse Events (participants affected / at risk) | 9/9 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MRKAd5 HIV-1 Gag Vaccine 1x10^9 vp/Dose (N=9) | Placebo (N=8)
Hepatitis C (Infections and infestations) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MRKAd5 HIV-1 Gag Vaccine 1x10^9 vp/Dose (N=9) | Placebo (N=8)
Palpitations (Cardiac disorders) | 1 | 0
Eye oedema (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 2 | 1
Fatigue (General disorders) | 1 | 1
Feeling hot (General disorders) | 1 | 0
Injection Site Erythema (General disorders) | 2 | 0
Injection Site Pain (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 3 | 1
Thirst (General disorders) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 1
Sciatica (Nervous system disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1
Dependence (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
An interim analysis of a related study, V520 Protocol 023 (NCT00095576), showed that the MRKAd5 vaccine used in Protocol 022 (NCT00857311) was not efficacious; therefore, only a high level summary of the safety data was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As this study is part of a multicenter trial, publications derived from this study should include input from the principal investigator, his/her colleagues, the other investigators in this trial, and SPONSOR personnel.

The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. SPONSOR review can be expedited to meet publication guidelines.